CLINICAL TRIAL: NCT05004571
Title: A Randomized, Placebo-Controlled, Double-Blinded Single and Multiple Ascending Dose (SAD and MAD) Study of the Safety, Tolerability, and Pharmacokinetics of EQU-001 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of EQU-001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Equilibre Biopharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQU-101
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Safety Issues
Keywords: Healthy; Adult; Volunteer

STUDY DESIGN:
Intervention Model Description: 3:1 treatment to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo control 10 mg capsules or 20 mg capsules totaling 20 mg, 40 mg, 80 mg, or 120 mg will be given once orally to placebo subjects in the SAD portion of the study.
  10 mg capsules or 20 mg capsules totaling 20 mg, 40 mg, 80 mg, or 120 mg will be given once daily for 14 days orally to placebo subjects in the SAD portion of the study.
  Interventions: Drug: Placebo
- Study drug EQU-001 (Experimental): 10 mg capsules or 20 mg EQU-001 capsules totaling 20 mg, 40 mg, 80 mg, or 120 mg will be given once orally to active-treatment subjects in the SAD portion of the study.
  10 mg capsules or 20 mg EQU-001 capsules totaling 20 mg, 40 mg, 80 mg, or 120 mg will be given once daily for 14 days orally to active treatment subjects in the SAD portion of the study.
  Interventions: Drug: EQU-001

INTERVENTIONS:
Drug: EQU-001 — EQU-001 in 10 and 20 mg capsules
  Arms: Study drug EQU-001
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blinded single and multiple ascending dose (SAD and MAD) study of the safety, tolerability, and pharmacokinetics of EQU-001 in healthy volunteers.

DETAILED DESCRIPTION:
EQU-001 is a Phase 1 randomized, placebo-controlled, double-blind SAD/MAD study to evaluate safety, tolerability, PK, and high-fat food effects on EQU-001. Eight healthy adult participants will be enrolled in each of up to 5 cohorts in both the SAD and MAD portions of the study (10 mg, 20 mg, 40 mg, 80 mg, and 120 mg). The participants will be randomized 3:1, drug to placebo. The MAD dosing is for 14 days, to include a period of time where the study drug will be at steady-state. Eight participants from the SAD study (the 40 mg dose cohort or the MTD dose cohort, whichever dose is lower) will also complete a fed portion of the study.

This study of EQU-001 will provide baseline safety, tolerability, PK, and food effect data in healthy individuals and aims to identify drug-specific DLTs and an MTD. The PK component will characterize the PK of EQU-001 to inform dosing and may help to correlate exposures with any DLTs or other treatment-related AEs. The food effect component will characterize the effect of a high-fat meal on EQU-001 kinetics and exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years of age
2. Weight 60 kg to 90 kg
3. Willing and able to

   * communicate in English or Spanish
   * provide written informed consent to take part in the study
   * be available for all visits and able and willing to comply with all study procedural requirements
4. In general good health in the opinion of the investigator as defined by:

   1. The absence of clinically significant illness or surgery within 4 weeks of dosing. Participants vomiting within 24 hours before the first study drug administration will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator or designee.
   2. The absence of clinically significant neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease including uncontrolled diabetes.
5. Agree not to participate in other concurrent interventional and/or drug trials
6. Agree not to use nicotine containing products
7. Agree not to eat grapefruit, drink grapefruit juice or take St. John's wort for 5 days prior to study drug dosing and throughout the study.
8. If you or your heterosexual partner is pre-menopausal, you must agree to use an effective method of contraception and to continue use of an effective method for the duration of study participation and 2 weeks after. For this study, a clinical history of amenorrhea for ≥1 year without a separate identifiable cause and a medical history consistent with menopause meets criteria for post-menopausal. Acceptable methods are:

   * condom use together with an additional barrier method plus spermicide, hormonal methods, or an IUD
   * sterilization of participant or partner
   * heterosexual abstinence

Exclusion Criteria:

1. Pregnant or lactating
2. History of hypersensitivity to the EQU-001 API
3. History of EQU-001 API use within the previous 2 weeks
4. History of ocular conditions that interfere with pupillometry including inability to focus on an object 3 meters in front of them, current eye disorder under the care of an ophthalmologist, or pupil not readily distinguishable from the iris
5. History of excessive caffeine use (>8 cups of coffee or caffeine-containing energy drinks per day)
6. History of smoking or vaping within the past 3 months
7. History of substance abuse within 6 months (with the exception of medically indicated marijuana), including alcohol
8. Use of concomitant prescription medications within 5 days of the study drug dose
9. Use of an investigational drug or device or participation in an investigational study within 30 days prior to enrollment
10. Donation of blood within the previous 4 weeks
11. Has any of the following laboratory abnormalities at screening or baseline:

    1. Breathalyzer result ≥ 0.1
    2. Positive COVID test
    3. Positive urine drug screen
    4. Positive urine cotinine screen
    5. Total bilirubin or higher ≥ 1.5 x the site laboratory ULN
    6. ALT or ALT ≥ 2 x the site laboratory ULN
    7. HbA1c ≥ 6.5%
    8. Positive hCG (female pre-menopausal participants)
12. Received a COVID-19 vaccine within 7 days of the baseline visit
13. Any reason which, in the opinion of the PI, would prevent the subject from participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
AEs Grade 2 or higher | Up to 19 days
  As defined by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0, November 2017
Change in pupil size from low light under high-light conditions between baseline and day 1 for part 1 (SAD) and day 14 for part 2 (MAD) | day 1 SAD; day 14 MAD

SECONDARY OUTCOMES:
Number of participants in each MAD cohort who discontinue the study drug because of study drug effects | Up to 14 days
EQU-001 drug concentration in blood | From pre-dose to 120 hours post dose in SAD and from pre-dose to 120 hours post the first and 14th doses in the MAD
Differences in EQU-001 drug concentrations in blood and in the parameters below under fasted as compared with fed conditions | From pre-dose to 120 hours post dose
Incidence of DLTs | up to 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy Melsaether, MD, Study Director — Equilibre Biopharmaceuticals B.V.
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: No